CLINICAL TRIAL: NCT01867463
Title: Double Blind Dose-Escalating Randomized Controlled Phase 1 Study in Malaria Exposed Adults of the Safety and Immunogenicity of Pfs25-EPA/ Alhydrogel, a Transmission Blocking Vaccine Against Plasmodium Falciparum in Bancoumana, Mali
Brief Title: Testing Pfs25-EPA/Alhydrogel as a Potential Malaria Transmission Blocking Vaccine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Malaria Research and Training Center, Bamako, Mali (Other)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 999913109; 13-I-N109
Record Dates: First submitted 2013-05-16; First posted 2013-06-04 (Estimated); Last update posted 2018-07-05 (Actual); Status verified 2016-12-19

CONDITIONS: Malaria
Keywords: Antigen; Ookinetes; Mosquito; Membrane; Assay
MeSH Terms: conditions — Malaria | interventions — Euvax-B; Meningococcal Vaccines

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- Group 1 (Experimental): Group 1: n=20, randomized to receive 16 g Pfs25-EPA/Alhydrogel (n=10) or the comparator (EuvaxB, n=10) on D0, D56
  Interventions: Biological: Pfs25-EPA/Alhydrogel; Biological: Euvax B
- Group 2 (Experimental): Group 2: n=30, randomized to receive 47 g Pfs25-EPA/Alhydrogel (n=15) or the comparator (EuvaxB and Menactra , n=15) on D0, D56, D112, D480
  Interventions: Biological: Pfs25-EPA/Alhydrogel; Biological: Euvax B; Biological: Menactra
- Group 3 (Experimental): Group 3: n=70 randomized to receive 47 g Pfs25-EPA/Alhydrogel (n=35) or the comparator (EuvaxB and Menactra , n=35) on D0, D56, D112, D480
  Interventions: Biological: Pfs25-EPA/Alhydrogel; Biological: Euvax B; Biological: Menactra

INTERVENTIONS:
Biological: Pfs25-EPA/Alhydrogel — The Pfs25-EPA conjugate was produced by reaction between thiolated PpPfs25 and maleimideactivated EcEPA, followed by purification using size-exclusion chromatography. The cGMP Pfs25-EPA conjugate Lot# WRAIR1634 was manufactured at Walter Reed Bioproduction facility in cGMP compliance in May 2010. Alhydrogel (Brenntag, Denmark) is an aluminum hydroxide gel and has been extensively used as an adjuvant in licensed human vaccines. Alhydrogel is supplied as a sterile product in water without preservatives. Pfs25- EPA/Alhydrogel WRAIR Lot #1668 was manufactured and filled as single-use vials at Walter Reed Bioproduction facility in cGMP compliance in October 2010. Each vial contains 78 g/mL conjugated Pfs25, 93 g/mL conjugated EPA and 1600 g/mL Alhydrogel in a volume of 0.8 mL. The vial label reads: 78 g/mL Conjugated Pfs25 on Alhydrogel .
Biological: Euvax B — Euvax B consists of highly purified, noninfectious particles of HBsAg absorbed onto aluminum salts as an adjuvant and preserved with thimerosal.
Biological: Menactra — Menactra , Meningococcal (Groups A, C, Y and W-135) Polysaccharide Diphtheria Toxoid Conjugate Vaccine, is a sterile, intramuscularly administered vaccine that contains Neisseria meningitidis serogroup A, C, Y and W-135 capsular polysaccharide antigens individually conjugated to diphtheria toxoid protein. N meningitidis A, C, Y and W-135 strains are cultured on Mueller Hinton agar (3) and grown in Watson Scherp (4) media. The polysaccharides are extracted from the N meningitidis cells and purified by centrifugation, detergent precipitation, alcohol precipitation, solvent extraction and diafiltration.
  Arms: Group 2; Group 3

SUMMARY:
Background:

- Malaria is a disease that is spread by mosquitoes. Researchers are looking for a vaccine that can prevent mosquitoes from transmitting malaria to people. They want to test a vaccine called Pfs25-EPA/Alhydrogel that may help stop malaria parasites from developing in mosquitoes. When a mosquito bites a vaccinated person, the vaccine should prevent parasites from developing in the mosquito. As a result, the mosquito will not spread malaria to the next person it bites. However, the vaccine will not directly prevent people vaccinated from getting sick with malaria. Researchers want to test this vaccine in people who live in rural Mali. To do so, the study will compare the symptoms and the blood tests of the participants who receive either the study vaccine or a regular hepatitis B/meningococcal vaccine.

Objectives:

- To see if Pfs25-EPA/Alhydrogel is a safe and effective malaria vaccine.

Eligibility:

- Healthy volunteers between 18 and 45 years of age who live in Bancoumana, Mali.

Design:

* Participants will be screened with a medical history, physical exam, and blood tests.
* Participants will be separated into two groups. One group will have Pfs25-EPA/Alhydrogel to test the study vaccine. The other group will have the regular Hepatitis B vaccine series, meningococcal vaccine.
* In the study vaccine group, participants will have either a lower dose or a higher dose. For the lower dose, they will have two vaccine shots over 1 year. For the higher dose, they will have four vaccine shots over about 14 months.
* In the other vaccine group, participants will have the Hepatitis B vaccine series, meningococcal vaccine according to the standard dose schedule.
* All participants will provide regular blood samples for testing during the study.
* Participants who develop malaria during the study will participate in evaluation of transmission and parasite development of malaria parasite from the person to mosquito via transmission assays. They will allow mosquitoes (that have no diseases) to bite them in a controlled clinic setting. This will let researchers see if the vaccine can stop the mosquitoes from carrying malaria to other people.

DETAILED DESCRIPTION:
A vaccine to interrupt malaria transmission would be a valuable tool for local elimination or eradication of this disease. Pfs25, a surface antigen of ookinetes in the mosquito stage of P. falciparum, is a lead candidate for a malaria transmission blocking vaccine. Recombinant Pfs25 has been conjugated to Pseudomonas aeruginosa ExoProtein A (EPA), and adjuvanted with Alhydrogel . This dose escalating, double-blind, randomized controlled trial will determine safety and immunogenicity of the vaccine in malaria exposed adults. One hundred twenty (120) subjects will be enrolled and randomized to receive the low dose (16 g of conjugated Pfs25, n=10), the high dose (47 g of conjugated Pfs25, n=50), or the comparator vaccine (Euvax B for first 3 vaccinations, then Menactra vaccine for the fourth vaccination, n=10 for 2 vaccinations, n=50 for 4 vaccinations). Enrollment within the high dose group will be staggered for additional safety. The low dose and the matching comparator cohort (Group 1) will receive 2 vaccine doses given at 0 and 2 months. For the rest of the subjects, 3 doses will be given at a 0, 2, 4 month dosing intervals, and a fourth (booster) dose will be given 12 months following the third dose at the start of the subsequent transmission season. Subjects will be followed for 12 months following the last vaccination. Safety outcomes will be local and systemic adverse events (AEs) and serious adverse events (SAEs). Immunogenicity outcomes will be antibody responses as measured by ELISA against recombinant Pfs25 and EPA, and B cell responses. Functional activity of the induced antibody will be assessed by direct transmission blocking assays (direct skin feeds, direct membrane feeding assays) conducted at the Malaria Research and Training Center (MRTC) in Mali and in a standard membrane feeding assay conducted at the National Institute of Allergy and Infectious Diseases (NIAID) in the United States.

ELIGIBILITY:
* INCLUSION CRITERIA:

All of the following criteria must be fulfilled for a subject to participate in this trial:

1. Adult age 18 45 years.
2. Known residents of the village of Bancoumana or immediate surrounding areas.
3. Available for the duration of the trial (approximately 2.5 years).
4. Good general health as a result of review of medical history and/or clinical testing at the time of screening.
5. Willingness to participate in the study as evidenced by signing the informed consent document, or by fingerprinting the consent document with the signature of a witness.
6. Willingness to undergo a HIV test.
7. Willingness to undergo direct skin feeds.

EXCLUSION CRITERIA:

A subject will be excluded from participating in this trial if any one of the following criteria is fulfilled:

1. Pregnancy, as determined by a positive urine or serum human choriogonadotropin (beta human chorionic gonadotropin ) test at any point during the study (if female).
2. Currently lactating and breast-feeding (if female).
3. Unable or unwilling to use reliable contraception for a minimum of one month prior to the first vaccination to three months after the last vaccination (if female). Reliable birth control includes: pharmacologic contraceptives including oral, parenteral, and transcutaneous delivery; condoms with spermicide; diaphragm with spermicide; surgical sterilization; vaginal ring; transdermal patch; intrauterine device; abstinence; and postmenopause.

   (Note: If screening of the female subject occurs < 1 month prior to first vaccination, a negative serum pregnancy test at time of screening and at enrollment (first vaccination) and agreement to use of reliable contraception for the duration of the study until three months after the fourth vaccination is acceptable.)
4. Behavioral, cognitive, or psychiatric disease that in the opinion of the investigator affects the ability of the participant to understand and cooperate with the study protocol.
5. Hemoglobin, WBC, and platelets outside the local laboratory-defined upper limit of normal (subjects may be included at the investigator s discretion for not clinically significant values outside of normal range).
6. Neutropenia (absolute neutrophil count <1250/mm3).
7. Alanine transaminase (ALT) or creatinine (Cr) level above the local laboratory-defined upper limit of normal.
8. Positive test for hepatitis C virus (HCV).
9. Positive test for hepatitis B (HBsAg).
10. Positive test for human immunodeficiency virus (HIV).
11. Known immunodeficiency syndrome.
12. Evidence of clinically significant neurologic, cardiac, pulmonary, hepatic, endocrine, rheumatologic, autoimmune, hematological, or renal disease by history, physical examination, and/or laboratory studies including urinalysis.
13. Subject has had medical, occupational, or family problems as a result of alcohol or illicit drug use during the past 12 months.
14. History of a severe allergic reaction or anaphylaxis.
15. History of a severe reaction to mosquito bites.
16. Severe asthma, defined as asthma that is unstable or required emergent care, urgent care, hospitalization or intubation during the past 2 years, or that has required the use of oral or parenteral corticosteroids at any time during the past 2 years.
17. Clinically significant reactive airway disease that does not respond to bronchodilators.
18. History of a surgical splenectomy.
19. Use of chronic (greater than or equal to 14 days) oral or intravenous corticosteroids (excluding topical or nasal) at immunosuppressive doses (i.e., prednisone >10 mg/ day) or immunosuppressive drugs within 30 days of starting this study.
20. Receipt of a live vaccine within past four weeks or a killed vaccine within past two weeks prior to entry into the study.
21. Receipt of blood products within the past 6 months.
22. Previous participation in a malaria vaccine trial.
23. History of receiving any investigational product within the past 30 days.
24. Refusal to allow storage of samples for future research at the time of enrollment.
25. Any medical, psychiatric, social, or occupational condition that, in the judgment of the Principal Investigator (PI), would interfere with the evaluation of study objectives or increase risk to the subject.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 230 (Actual)
Dates: Start 2013-03-27; Primary Completion 2015-12-22 (Actual); Study Completion 2016-12-19 (Actual)

PRIMARY OUTCOMES:
Incidence of local and systemic adverse events and serious adverse events. | 12 months following the last vaccination; and for 6 months following the fourth vaccination.

SECONDARY OUTCOMES:
Antibody responses as measured by ELISA against recombinant Pfs25 and EPA, and B cell responses. Functional activity of the induced antibody will be assessed by direct transmission blocking assays | 12 months following the last vaccination; and for 6 months following the fourth vaccination.

CONTACTS AND LOCATIONS:
Overall Officials: Sara A Healy, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- Malaria Research and Training Center, Bamako, Mali

REFERENCES:
- [Background] Kaslow DC. Transmission-blocking vaccines. Chem Immunol. 2002;80:287-307. doi: 10.1159/000058850. No abstract available. PMID 12058646
- [Background] Williamson KC, Keister DB, Muratova O, Kaslow DC. Recombinant Pfs230, a Plasmodium falciparum gametocyte protein, induces antisera that reduce the infectivity of Plasmodium falciparum to mosquitoes. Mol Biochem Parasitol. 1995 Dec;75(1):33-42. doi: 10.1016/0166-6851(95)02507-3. PMID 8720173
- [Background] Diallo M, Toure AM, Traore SF, Niare O, Kassambara L, Konare A, Coulibaly M, Bagayogo M, Beier JC, Sakai RK, Toure YT, Doumbo OK. Evaluation and optimization of membrane feeding compared to direct feeding as an assay for infectivity. Malar J. 2008 Dec 2;7:248. doi: 10.1186/1475-2875-7-248. PMID 19055715
- [Derived] Sagara I, Healy SA, Assadou MH, Gabriel EE, Kone M, Sissoko K, Tembine I, Guindo MA, Doucoure M, Niare K, Dolo A, Rausch KM, Narum DL, Jones DL, MacDonald NJ, Zhu D, Mohan R, Muratova O, Baber I, Coulibaly MB, Fay MP, Anderson C, Wu Y, Traore SF, Doumbo OK, Duffy PE. Safety and immunogenicity of Pfs25H-EPA/Alhydrogel, a transmission-blocking vaccine against Plasmodium falciparum: a randomised, double-blind, comparator-controlled, dose-escalation study in healthy Malian adults. Lancet Infect Dis. 2018 Sep;18(9):969-982. doi: 10.1016/S1473-3099(18)30344-X. Epub 2018 Jul 27. PMID 30061051